CLINICAL TRIAL: NCT03351127
Title: The Multi-center Normal Reference Study of Carotid Artery Ultrafast Pulse Wave Velocity (UFPWV) in Chinese Han Adults (CAR-PWV Study）
Brief Title: Multicenter Normal Reference Study of Carotid Artery Ultrafast Pulse Wave Velocity (UFPWV)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shengjing Hospital (Other)
Collaborators: SuperSonic Imagine (Industry)
Responsible Party: Principal Investigator, Weidong Ren, Director of Ultrasonic Department, Shengjing Hospital
Other Study IDs: ShengjingH-RWD
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Carotid Artery Diseases; Healthy Volunteers
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 18-29 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 18-29 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination
- 30-39 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 30-39 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination
- 40-49 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 40-49 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination
- 50-59 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 50-59 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination
- 60-69 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 60-69 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination
- 70-79 year-old group: Based on the inclusion crtiteria, 200 healthy Han people at aged 70-79 and both sexes will be recruited in the analysis. Normal reference values of ultrafast pulse wave velocity will be obtained.
  Interventions: Radiation: Carotid ultrasound examination

INTERVENTIONS:
Radiation: Carotid ultrasound examination — Carotid pulse wave velocity of all participants were measured by ultrafast ultrasound imaging technology using SuperSonic Imagine's Aixplorer ultrasound system.

SUMMARY:
To establish the range of BS and ES (m/s) of normal carotid artery by using ultrafast pulse wave velocity (UFPWV), and to explore the influencing factors.

DETAILED DESCRIPTION:
With the gradual aging of Chinese population and continuous development of economy and society, the incidence of cardiovascular disease and the number of patients have increased rapidly. The National Heart Center has reported that the number of patients with clinically diagnosed cardiovascular disease in China has reached 290 million in 2016 (240 million in 2014). Cardiovascular disease is the most common cause of death in humans, accounting for nearly 60% of all deaths worldwide. The updated data from World Health Organization (WHO) in 2008 have shown that atherosclerosis and hypertension are the major diseases of the cardiovascular system. Therefore, early detection of arteriosclerosis, timely treatment and early evaluation of therapeutic efficacy are of great significance for the overall control and reduction of the incidence and mortality of cardiovascular disease.

Carotid artery intima-media thickness (IMT) is often used to evaluate early atherosclerosis, but IMT reflects the change of vascular wall structure. In the early stage of atherosclerosis, the changes of vascular elasticity and resistance occur earlier than those of arterial wall thickening. Therefore, accurate evaluation of vascular function plays an important role in the early diagnosis of atherosclerosis.

Basic and clinical studies and clinical data have shown that pulse wave velocity (PWV) is a reliable index for early evaluation of atherosclerosis. The blood is pumped from the left ventricle during systole, and travels along the arterial system to form pulse wave. Its propagation velocity between two fixed points is the PWV. Atherosclerosis leads to the increased PWV. The detection of PWV can accurately reflect the distensibility and stiffness of arterial wall, thereby early detecting atherosclerosis.

There are three main methods for non-invasive pulse wave measurement: Photoelectric sensor is used to measure and record photoplethysmography signal. Pressure sensor is utilized to record pressure wave signals produced by arterial pulsation on the body surface. Ultrasonic Doppler sensor is applied to collect photoplethysmography signal. Photoelectric sensor acquisition system is difficult to distinguish the pulse waves between the large artery and the capillary arteriole, cannot detect the signal of the deep aorta, is easily affected by the electrical signals of perivascular tissue, and has not been widely used in the clinic. Pressure sensor can be used to collect pressure wave signals, such as brachial-ankle pulse wave. This method has relatively low cost, is often used in clinic, but cannot directly get the pulse wave form and the distance of blood vessel, has many influencing factors and low accuracy. Ultrasonic Doppler technique, such as Echo Tracking and QSA, can reveal deep vein pulse waveforms. However, limited by the traditional ultrasonic processing platform, signal acquisition and formula calculation are complex, and the repeatability is poor. Therefore, the clinical application value is limited. It is urgent to establish a new, simple and precise method for the detection of PWV.

ELIGIBILITY:
Inclusion Criteria:

* Han nationality
* Age between 18 and 79 years old
* Normal body mass index (18-25 kg/m2)
* Normal blood pressure (139-90/89-60 mmHg)
* No history of cardiovascular disease or respiratory diseases
* Physical examination reveals no abnormalities in cardiovascular and respiratory systems
* Normal blood glucose, blood lipid and electrocardiogram (ECG)
* Echocardiography shows no structural heart disease and normal cardiac function
* Normal carotid ultrasound
* No history of cardiovascular drug use

Exclusion Criteria:

* Heart valve regurgitation with clinical significance or moderate symptom and above
* Respiratory system disease: acute or chronic respiratory disease
* Endocrine diseases: thyroid disease, diabetes mellitus, aldosteronism, pheochromocytoma, and adrenal cortex dysfunction.
* Metabolic syndrome
* Anemia
* Pregnant or lactating women
* Abnormal liver function (more than twice the normal upper limit), abnormal renal function (creatinine > 2 mg/dl), total cholesterol > 190 mg/dl. If Pro-BNP is detected, Pro-BNP is abnormal or in high limit of normal value.
* Connective tissue disease
* Tumor
* Aortic and peripheral vascular diseases: aortic dilatation, aortic dissection, coarctation of the aorta, polyarteritis, atherosclerosis
* Daily drinking: liquor greater than 50 ml; red wine more than 100 ml; beer more than 300 ml
* Professional sportsman
* The poor quality of ultrasonic images cannot meet parameter measurement and analysis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1200 healthy adults with normal physical examination items will be selected from the physical examination center.
  According to sex and age stratification, totally 1200 cases will contain 600 males and 600 females.
  From 18 to 79 years old, they will be divided into 6 groups: 18-29 years, 30-39 years, 40-49 years, 50-59 years, 60-69 years and 70-79 years (n=200 per group).
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid pulse wave velocity at the beginning and end of systole | 1 day
  To establish the range of pulse wave velocity at the beginning of the systole (BS) and at the ending of the systole (ES) of normal carotid artery, and to identify the influencing factors for BS and ES in the carotid artery.

SECONDARY OUTCOMES:
Carotid artery intima-media thickness (IMT) | 1 day
  IMT reflects the change of vascular wall structure, which is used to evaluate early atherosclerosis and .
Serum biochemical index | 1 day
  Serum laboratory testing for blood cholesterol level (total cholesterol, HDL (high-density lipoprotein), LDL (low-density lipoproteins), triglycerides), fasting blood-glucose will be examed.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Ren, Principal Investigator — Shengjing Hospital of China Medical Univeristy; Lixue Yin, Principal Investigator — People's Hospital of Sichuan Province
Locations (44):
- China (44):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Civil Aviation General Hospital, Beijing, Beijing Municipality
  - University-Town Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Central Hospital of Chongqing Three Gorges, Chongqing, Chongqing Municipality
  - Guangdong Second Traditional Chinese Medicine Hospital, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Huadu District People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of He'nan University of Science and Technology, Luoyang, He'nan
  - The First People's Hospital of Pingdingshan of He'nan Province, Pingdingshan, He'nan
  - Xinxiang Central Hospital, Xinxiang, He'nan
  - Zhengzhou Tumor Hospital Affiliated to He'nan University, Zhengzhou, He'nan
  - He'nan Provincial People's Hospital, Zhengzhou, He'nan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, He'nan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, He'nan
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The Second Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Wuchang Hospital of Hubei Province, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Province Hospital of Traditional Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Provincial Geriatric Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Central Hospital Affiliated to Shenyang Medical College, Shenyang, Liaoning
  - The First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Yan'an University Affiliated Hospital, Yan’an, Shanxi
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The First Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Xinjiang Uygur Autonomous Region Hospital of Traditional Chinese Medicine, Ürümqi, Xinjiang
  - Hangzhou Hospital of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang